CLINICAL TRIAL: NCT00680446
Title: An Open-Label Study of Ig NextGen 16% Administered by Subcutaneous Infusion in Patients With Primary Immunodeficiency (PID).
Brief Title: Safety Study of Subcutaneous Ig NextGen 16% in Patients With Primary Immunodeficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CSL Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSLCT-SCIG-07-42
Record Dates: First submitted 2008-05-16; First posted 2008-05-20 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Primary Immune Deficiency
Keywords: Primary Immune Deficiency; Subcutaneous; Immunoglobulin G
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Immunoglobulin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Immunoglobulin G (Ig NextGen 16%)

INTERVENTIONS:
Drug: Immunoglobulin G (Ig NextGen 16%) — Weekly or Bi-weekly subcutaneous administration of Immunoglobulin G
  Other Names: Ig NextGen 16%

SUMMARY:
The study aims to assess the safety and tolerability of subcutaneous Ig NextGen 16% in patients with Primary Immune Deficiency who require Immunoglobulin (Ig) G replacement therapy. Ig NextGen 16% is a liquid immunoglobulin (antibody) preparation.

DETAILED DESCRIPTION:
This is a Phase 3, open label, multi-centre, study for patients requiring Ig replacement therapy. This study is a follow-on study to patients who have completed the CSLCT-SCIG-05-23 clinical trial and wish to continue subcutaneous treatment with Ig NextGen 16% . Additionally, patients currently receiving IVIg with unacceptable adverse reactions or unable to tolerate IVIg as well as patients receiving alternate IG products via the SC route may be enrolled in this study. Patients must not be eligible for any of the Sponsor's ongoing PID studies that are still open to enrolment.

ELIGIBILITY:
Inclusion Criteria:

1. Age >3 years of age.
2. PID patients receiving Ig replacement therapy.
3. Patients must have completed or withdrawn from CSLCT-SCIG-05-23 and wish to continue SCIg therapy; or, patients ineligible for CSLCT-SCIG-05-23 but for whom the Investigator believes SCIg may be a suitable form of Ig replacement, for reasons such as: poor tolerability of IVIg, difficult venous access, or, preferred route of administration.
4. Patient is capable of self-administering Ig NextGen 16%

Exclusion Criteria:

1. Patients eligible for CSLCT-SCIG-05-23 if still open for recruitment.
2. Patients with known anaphylaxis reactions to immunoglobulin therapy.
3. Patients with known selective IgA deficiency or antibodies to IgA with a history of reactions to Ig therapy.
4. Patients with protein-losing enteropathies.
5. Patients who are suffering from an acute or chronic medical condition, other than PID, which may, in the opinion of the Investigator, affect their treatment or the conduct of the trial.
6. Females who are pregnant, breast feeding or planning a pregnancy during the course of the study. Females who are of child bearing potential must have a negative pregnancy test at screening.
7. Patients unwilling to comply with the protocol.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Rate, Severity and Relatedness of reported Adverse Events | Up to Four Years

SECONDARY OUTCOMES:
To monitor patient IgG trough levels while receiving Ig NextGen 16% | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical and Research Director, Study Director — CSL
Locations (9):
- Australia (6):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - Sydney Children's Hospital, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Women's & Children's Hospital, North Adelaide, South Australia
  - Frankston Hospital, Frankston, Victoria
  - Royal Children's Hospital, Parkville, Victoria
- New Zealand (3):
  - Auckland Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Wellington Hospital, Wellington